CLINICAL TRIAL: NCT00589836
Title: Assessment of LV Torsion by Tissue Doppler Echocardiography
Brief Title: Assessment of Left Ventricular Torsion by Echocardiography Study
Acronym: LVTorsion
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Zoran Popovic, Principal Investigator, The Cleveland Clinic
Other Study IDs: IRB 05-023
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Results first posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2017-07

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: HCM; HOCM; hypertrophic cardiomyopathy; tissue doppler echocardiography; myocardial torsion
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Pathologies: Patients with cardiomyopathy, ischemic heart disease, will have tissue Doppler echocardiograms performed

SUMMARY:
The purpose of this study is to learn about the twisting or wringing motion of the heartbeat called Left Ventricular Torsion (LV Torsion) which can be seen on ultrasound.

DETAILED DESCRIPTION:
This study is designed to characterize the myocardial torsional behavior in patients with a variety of cardiac pathologies.

Simple and inexpensive methods for measurement of LV torsion could facilitate more widespread investigation of LV torsion, which might reveal significant relationships between torsional alterations and clinical outcomes and eventually lead to routine clinical application. Recently, Doppler tissue imaging (DTI) has been shown to accurately reflect myocardial velocity24,25 with better temporal resolution than MRI.26 Investigators hypothesize therefore that DTI might be used for quantification of LV rotation and torsion of the human heart. The purpose of the present study was to examine the accuracy of a novel method with DTI for quantifying the LV torsion in humans and tagged MRI as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age 18 to 70 years
* Patients with hypertrophic cardiomyopathy
* Patients with the ability to exercise using a supine bicycle
* Ability to provide informed consent

Exclusion Criteria:

* Aortic valve stenosis classified as moderate to severe
* Severe left ventricular obstruction at rest (high gradients > 4m/second)
* Uncontrolled arrhythmias including atrial fibrillation, atrial flutter, frequent premature ventricular ectopic beats
* History of sustained ventricular tachyarrhythmia at any time

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac echocardiography testing in the outpatient department
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2005-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zoran Popovic, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Consecutive patients with clinically indicated MRI and previous satisfactory echocardiographic images on a previously performed study had a research echocardiographic study on the same day as the MRI
Groups:
- Cardiac Pathologies: Clinical diagnosis included aortic root disorder, severe aortic insufficiency, severe aortic stenosis, post aortic valve replacement, and cardiomyopathies.
Period: Overall Study
Arm/Group | Cardiac Pathologies
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Cardiac Pathologies: Patients with cardiac pathologies of aortic root disorder, severe aortic stenosis, severe aortic insufficiency, aortic valve replacement, ischemic heart disease and cardiomyopathies had tissue DTI and MRI performed
Arm/Group | Cardiac Pathologies
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Doppler Tissue Imaging
Description: The purpose of the present study was to examine the accuracy of a novel method with DTI for quantifying the LV torsion in humans and tagged MRI as the reference standard.
  LV torsion reflects the torsion (twisting deformation) occurring across the length of the ventricle (from the base to the apex) during the time interval defined by the beginning and end of contraction (or in physiologic terms, from end -diastole to end systole). In this study, end diastole was defined by the R wave of the ECG, while end systole is defined by minimum end-systolic volume or maximum of twisting deformation. The deformation is measured in degrees.
  Once the measurements are performed by experimental method (i.e. TDI imaging) and reference method (i.e. MRI imaging) these two methods are then compared using Bland Altman analysis.
  In a current study, mean difference between methods of torsion quantification was 0.57 degrees, while the standard deviation (SD) was 1.98 degrees.
Time Frame: 1 1/2 hours
Population: population had both MRI and DTI on the same day.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Cardiac Pathologies
Number analyzed (Participants) | 20
degrees | 0.57 (1.98)

ADVERSE EVENTS:
Time Frame: 1.5 Hours
Arm/Group | Cardiac Pathologies
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes